CLINICAL TRIAL: NCT01081249
Title: Physiologic Correlates of Perceived [Therapist] Empathy and Social-Emotional Process During Psychotherapy: Testing Oxytocin in a Cross-Over Design Pilot Study
Brief Title: Effects of Oxytocin on Behavior and Physiology in a Psychotherapy Setting
Acronym: OT-PT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MacDonald, Kai, M.D. (Individual)
Responsible Party: Principal Investigator, Kai MacDonald, Assistant clinical professor, MacDonald, Kai, M.D.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD IRB 080953
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Behavior; Anxiety
Keywords: psychotherapy
MeSH Terms: conditions — Behavior; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then Oxytocin (Experimental): Participant was randomized to receive placebo before the first psychotherapy session, and then received the active drug at the second visit.
  Interventions: Drug: Placebo then intranasal oxytocin
- Oxytocin then placebo (Experimental): Participant was randomized to receive placebo before the first psychotherapy session, and then received the active drug at the second visit.
  Interventions: Drug: Intranasal oxytocin then placebo

INTERVENTIONS:
Drug: Placebo then intranasal oxytocin — Participant received intranasal placebo spray at first psychotherapy session, and received a single dose of 40 IU intranasal oxytocin at the second session.
  Arms: Placebo then Oxytocin
Drug: Intranasal oxytocin then placebo — Participant received a single dose of 40 IU intranasal oxytocin at the first psychotherapy session, and received a similar dose of intranasal placebo spray at the second session.
  Arms: Oxytocin then placebo

SUMMARY:
Subjects-currently in outpatient mental health care--will participate in 2 psychotherapy sessions, one with oxytocin spray and one with placebo spray. Sessions will be videotaped, and cortisol and heart rate will be measured. We hypothesize that oxytocin will have positive benefits on nonverbal behavior in the therapy session, as well as have positive effects on subjective anxiety, cortisol and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* in current mental health treatment
* male 18-65

Exclusion Criteria:

* diagnosis of schizophrenia or psychosis
* diagnosis of autism or Aspergers disorder
* active substance use disorder
* at moderate or high risk of self-harm

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai MacDonald, MD, Principal Investigator — UCSD
Locations (1):
- Kai MacDonald, MD 3368 2nd Ave Ste B, San Diego, California, United States

REFERENCES:
- [Background] Macdonald K, Macdonald TM. The peptide that binds: a systematic review of oxytocin and its prosocial effects in humans. Harv Rev Psychiatry. 2010 Jan-Feb;18(1):1-21. doi: 10.3109/10673220903523615. PMID 20047458
- [Derived] MacDonald K, MacDonald TM, Brune M, Lamb K, Wilson MP, Golshan S, Feifel D. Oxytocin and psychotherapy: a pilot study of its physiological, behavioral and subjective effects in males with depression. Psychoneuroendocrinology. 2013 Dec;38(12):2831-43. doi: 10.1016/j.psyneuen.2013.05.014. Epub 2013 Jun 28. PMID 23810433

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin Then Placebo: Participants received a single dose of 40 IU intranasal oxytocin prior to the first psychotherapy session; prior to the second psychotherapy session they received a similar dose of intranasal placebo.
- Placebo Then Oxytocin: Participants received a single dose of intranasal placebo prior to the first psychotherapy session; prior to the second psychotherapy session the participants received a single dose of 40 IU intranasal oxytocin.
Period: Overall Study
Arm/Group | Oxytocin Then Placebo | Placebo Then Oxytocin
Started | 11 | 7
First Psychotherapy Appointment (1 Day) | 11 | 6
Washout (5-10 Days) | 11 | 6
Second Psychotherapy Appointment (1 Day) | 11 | 6
Completed | 11 | 6
Not Completed | 0 | 1
Not completed — Diagnosed with Bipolar Disorder | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Drug: placebo
  intranasal oxytocin: single dose of 40 IU intranasal oxytocin or similar volume of placebo
  placebo: single dose of 40 IU intranasal oxytocin or similar volume of placebo
Arm/Group | Active Drug
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Verbal and Nonverbal Behavior in Therapy Session: Effects of Drug
Description: Videotapes of 2 therapy session (PBO/OT) were reviewed by blinded raters to determine differences in two treatments. There were nine aspects analyzed using the Ethological Coding System for Interviews: eye contact, affiliation, submission, prosocial, flight, assertion, displacement, relaxation, and gesture.
Time Frame: videotapes of session were reviewed and scored 1-3 months after the patient completes the study
Measure: Mean (Standard Deviation); unit: Number of behaviors exhibited
Groups:
- Placebo: A dose of intranasal placebo was administered prior to the psychotherapy session.
- Active Drug: A dose of 40 IU intranasal oxytocin was administered prior to the psychotherapy session.
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 17 | 17
Number of behaviors exhibited
  ECSI eye contact | 34 (2.2) | 34.8 (2.4)
  ECSI affiliation | 45.4 (5.1) | 46.0 (4.5)
  ECSI submission | 24.4 (6.1) | 25.14 (5.6)
  ECSI prosocial | 69.8 (7.3) | 71.1 (7.3)
  ECSI flight | 65.7 (2.9) | 61.1 (4.0)
  ECSI assertion | 30.5 (5.7) | 26.6 (3.9)
  ECSI displacement | 46.6 (3.9) | 41.6 (5.2)
  ECSI relaxation | 19.4 (4.4) | 18.7 (3.3)
  ECSI gesture | 28.8 (3.0) | 29.3 (2.2)

2. Secondary Outcome: Salivary Cortisol
Description: Salivary cortisol will be measured after the treatment, and before, during and after the therapy session.
Time Frame: before drug, before session, and 20 minutes after session
Reporting Status: Not Posted

3. Secondary Outcome: Heart Rate Variability (HRV)
Description: HRV will be measured before, during and after the therapy session.
Time Frame: continuously monitored from time before drug delivery to 20 minutes after session
Reporting Status: Not Posted

4. Secondary Outcome: Subjective Ratings of Anxiety and Trust of the Therapist
Description: Patient will fill out ratings of subjective anxiety (STAI), mood and energy (PANAS), and trust (Likert scale) in the therapist before and after the session.
Time Frame: measured before drug, immediately before session, and after the session
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Placebo Then Oxytocin: Participants received intranasal placebo spray prior to the first psychotherapy session; prior to the second psychotherapy session they received 40 IU intranasal oxytocin.
- Oxytocin Then Placebo: Participants received 40 IU intranasal oxytocin prior to the first psychotherapy session; prior to the second psychotherapy session they received a comparable dose of intranasal placebo spray.
Arm/Group | Placebo Then Oxytocin | Oxytocin Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 0/6 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No